CLINICAL TRIAL: NCT03506802
Title: Adoptive Transfer of NY-ESO-1 TCR Engineered Peripheral Blood Mononuclear Cells (PBMC) and Peripheral Blood Stem Cells (PBSC) After a High Dose Melphalan Conditioning Regimen, With Administration of Interleukin-2, in Patients With Multiple Myeloma
Brief Title: TCR Genetically Engineered PBMC and PBSC After Melphalan Conditioning Regimen in Treating Participants With Relapsed and Refractory Multiple Myeloma
Acronym: NYSCT MM
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001866; NCI-2018-00204 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-001866 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-06

CONDITIONS: HLA-A*0201 Positive Cells Present; NY-ESO-1 Positive Tumor Cells Present; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 9-(4-fluoro-3-hydroxymethylbutyl)guanine; aldesleukin; Cell- and Tissue-Based Therapy; Filgrastim; Granulocyte Colony-Stimulating Factor; Lenalidomide; Leukapheresis; Melphalan; plerixafor; ferric pyrophosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Genetically engineered PBMC and PBSC) (Experimental): Refer to outline
  Interventions: Radiation: 18F-FHBG; Biological: Aldesleukin; Biological: Cellular Therapy; Procedure: Computed Tomography; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Procedure: Leukapheresis; Drug: Melphalan; Drug: Plerixafor; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: 18F-FHBG — Given IV
  Other Names: Reporter Probe 18F-FHBG
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Cellular Therapy — LV-NYESO TCR /sr39TK PBSC and RV-NYESO TCR PBMC given IV
  Other Names: Cell Therapy
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies the side effects of NY-ESO-1 TCR engineered peripheral blood mononuclear cells (PBMC) and peripheral blood stem cells (PBSC) after melphalan conditioning regimen in treating participants with multiple myeloma that has come back or does not respond to treatment. The melphalan conditioning chemotherapy makes room in the patient?s bone marrow for new blood cells (PBMC) and blood-forming cells (stem cells) to grow. Giving NY-ESO-1 TCR PBMC and stem cells after the conditioning chemotherapy is intended to replace the immune system with new immune cells that have been redirected to attack and kill the cancer cells and thereby improve immune system function against cancer. Giving NY-ESO-1 TCR PBMC and PBSC after melphalan may work better at treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of administering the combination of autologous peripheral blood mononuclear cells (PBMC) and CD34+ peripheral blood stem cells (PBSC) following a melphalan conditioning regimen, both of which have been genetically modified to express NY-ESO-1 TCR.

SECONDARY OBJECTIVES:

I. To determine the feasibility of delivering the combination of T-cell receptor (TCR) transduced autologous PBMC and CD34+ PBSC to patients.

II. To determine the persistence of NY-ESO-1 TCR transduced PBMC and the progeny of TCR transduced PBSC in serial peripheral blood samples.

III. Objective response rate (ORR).

TERTIARY OBJECTIVES:

I. To explore the use of positron emission tomography (PET)-based imaging using the PET tracer 9-4-[18F]fluoro-3-(hydroxymethyl)butylguanine ([18F]FHBG) with the goal of determining whether the adoptively transferred NY-ESO-1 TCR transduced PBSC home to bone marrow, differentiate into T cells and expand in secondary lymphoid organs and extramedullary disease sites.

OUTLINE:

G-CSF AND PLERIXAFOR MOBILIZED LEUKAPHERESIS: Between 6 months and 3 weeks before infusion of cells, participants undergo G-CSF and plerixafor mobilization of CD34+ peripheral blood stem cells. Participants receive filgrastim subcutaneously (SC) on mobilization days 1-4 and up to mobilization day 8 and plerixafor SC starting on mobilization day 4 up to day 8. During mobilization, participants will undergo mobilized leukapheresis to obtain PBSC. Participants also undergo an unmobilized leukapheresis on day -5 before infusion of cells in order to obtain PBMC.

CHEMOTHERAPY CONDITIONING REGIMEN: Participants receive melphalan intravenously (IV) on days -3 to -2.

Participants receive LV-NYESO TCR/sr39TK PBSC IV on day 0, and RV-NYESO TCR PBMC IV on day 1. Beginning on day 2, participants receive aldesleukin (interleukin-2 or IL-2) SC twice daily (BID) for up to 7 days. Participants receive the 18F-FHBG IV, and after 1 hour, undergo PET/computed tomography (CT) on days 30 and 90. After day 100, participants receive lenalidomide orally (PO) once daily (QD) for 21 days. Courses of lenalidomide repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up monthly after day 90 until disease progression and annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed, relapsed and refractory or refractory multiple myeloma patients who have received > 3 prior lines of therapy including a proteasome inhibitor, an immunomodulatory agent, and an anti-CD28 monoclonal antibody
* NY-ESO-1 positive by immunohistochemistry (IHC) utilizing commercially available NY-ESO-1 antibodies
* HLA-A*0201 (HLA-A2.1) positivity by molecular subtyping
* Measurable disease defined by at least one of the following:

  * Serum monoclonal protein (serum protein electrophoresis [SPEP]) > 1gm/dL
  * Serum free light chain (sFLC): involved free light chain (FLC) >= 10mg/dL AND abnormal kappa to lambda serum free light chain ratio
  * >= 200mg of monoclonal protein in the urine on 24 hour electrophoresis (urine protein electrophoresis [UPEP])
* Adequate bone marrow and major organ function to undergo a PBSC transplant determined within 30-60 days prior to enrollment using standard phase 1 criteria for organ function defined as:

  * Absolute neutrophil count (ANC) >= 1.5 x 10^9 cells/L
  * Platelets >= 75 x 10^9/L
  * Hemoglobin >= 8 g/dL
  * Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN, if documented liver metastases are present)
  * Total bilirubin =< 2 x ULN (except patients with documented Gilbert?s syndrome)
  * Creatinine < 2 mg/dl (or a glomerular filtration rate > 60)
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Must be willing and able to accept at least three leukapheresis procedures
* Must be willing and able to undergo three research PET scans
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Inability to purify >= 2.5 x 10^6 CD34-enriched cells/kg of patient weight from the pooled granulocyte-colony stimulating factor (G-CSF) mobilized leukapheresis products
* Previous allogeneic transplant
* Previously known hypersensitivity to any of the agents used in this study; known sensitivity to melphalan
* Received systemic treatment for multiple myeloma, including immunotherapy, within 14 days prior to initiation of study procedures
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Known clinically active central nervous system (CNS) involvement; prior evidence of CNS involvement successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment and there are no neurological signs of potential CNS involvement
* Pregnancy or breast-feeding; female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and for 6 months afterwards; all female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 14 days from starting the conditioning chemotherapy; the definition of effective contraception will be based on the judgment of the study investigators
* Since IL-2 is administered following cell infusion:

  * Patients will be excluded if they have a history of clinically significant electrocardiogram (ECG) abnormalities, symptoms of cardiac ischemia with evidence of ischemia on a cardiac stress test (stress thallium, stress multigated acquisition [MUGA], dobutamine echocardiogram or other stress test)
  * Similarly, patients with a baseline left ventricular ejection fraction (LVEF) < 45 percent (%) will be excluded
  * Patients with ECG results of any conduction delays (PR interval > 200 ms, corrected QT [QTC] > 480 ms), sinus bradycardia (resting heart rate < 50 beats per minute), sinus tachycardia (heart rate > 120 beats per minute) will be evaluated by a cardiologist prior to starting the trial; patients with any arrhythmias, including atrial fibrillation/atrial flutter, excessive ectopy (defined as > 20 premature ventricular contractions [PVCs] per minute), ventricular tachycardia or 3rd degree heart block will be excluded from the study unless cleared by a cardiologist
  * Patients with pulmonary function test abnormalities as evidenced by a forced expiratory volume in 1 (FEV1) / forced vital capacity (FVC) < 70% of predicted for normality will be excluded
* Active or recent herpes simplex virus (HSV) infection or cytomegalovirus (CMV) based on symptoms with positive swab culture and/or positive Immunoglobulin M (IgM) screening, which would complicate the post-conditioning period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-06-25 (Estimated); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | Up to 90 days
  Safety will be assessed by monitoring and recording potential adverse effects of the treatment using the Common Toxicity Criteria at each study visit. Subjects will be monitored by medical histories, physical examinations and blood studies to detect potential toxicities from the treatment. If there are no dose limiting toxicities observed, the cohort will be expanded to 12 subjects. If 1/3 are observed, up to 6 subjects will be recruited. If less than 2/6 are observed, the cohort will be expanded to a total of 12 subjects. If a dose limiting toxicity is observed in 2 or more of 6 subjects, then this dose level will have exceeded the 33% rate, and the study will be terminated.

SECONDARY OUTCOMES:
Feasibility of NY-ESO-1 TCR transgenic cells | Up to 1 month after transgenic cell adoptive transfer
  The feasibility of manufacturing will be assessed as the number of manufacturing products meeting the lot release criteria after an acceptable number of CD34+ cells have been obtained.
Persistence of transduced T cells | Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed using immune monitoring techniques. The number of days until the percentage of cells expressing both NYESO-1 TCR and CD3 drops below the baseline percentage.
Engraftment and persistence of transduced progeny T cells | Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed using immune monitoring techniques. The number of days until the vector copy number in the progeny T cells is undetectable.
Engraftment and persistence of transduced T cells and progeny T cells | Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed both using immune monitoring and molecular techniques. The number of days until the vector copy number in the T cells is undetectable.
Persistence of TCR gene transduced cells | Up to 15 years
  Will be assessed by semi quantitative deoxyribonucleic acid-polymerase chain reaction using primers specific for vector sequence.
Long term monitoring for replication competence of retrovirus (RCR) and lentivirus (RCL) | Up to 12 months post cell administration
  Will be assessed by polymerase chain reaction.
Immunological monitoring | Up to 15 years
  Will be assessed by NY-ESO-1126-157/MHC dextramer analysis. Functional assays like enzyme-linked immunosorbent assay, intracellular cytokine staining, and/or multicytokine array assays will complement the results. Immunological assays will be compared between 1) pre-infusion peripheral blood mononuclear cells and peripheral blood stem cells, 2) an aliquot of the engineered peripheral blood lymphocytes and stem cells at the time of infusion and 3) cells recovered from patients? peripheral blood after adoptive transfer.
Objective response | Up to 15 years
  Potential objective responses to this combinatorial immunotherapy will be recorded following International Myeloma Working Group (IMWG) Response Criteria.
Duration of overall complete response | From the time measurement criteria has been first met for complete response until the first date that recurrent or progressive disease is objectively documented, assessed up to 15 years
  Will evaluate duration of overall complete response.
Duration of overall response | From the time measurement criteria is met for complete response/partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 15 years
  Will evaluate duration of overall response.
Time to disease progression | Time from the date of cell infusion (day 0) to the date of progressive disease first documented, or death whichever occurs first, assessed up to 15 years
  Will evaluate length of time until disease progression.

OTHER OUTCOMES:
LV-NYESO TCR/sr39TK peripheral blood stem cell (PBSC) biodistribution (Regional uptake of 18F-FHBG within metastatic tumor sites and secondary lymphoid organs) | Day 30 and day 90
  Will be quantified by standardized uptake values normalized to the body weight of the patient. As an internal quality control, standardized uptake values will also be determined for several normal organs, such as muscle, liver and lungs. These measurements will allow us to identify technical problems in the standardized uptake value calculations, such as partially paravenous tracer administration. Findings from non-invasive positron emission tomography imaging will be compared with results from immune monitoring assays in blood samples at different intervals after NY-ESO-1 TCR cell transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Larson, M.D., Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States